CLINICAL TRIAL: NCT02608775
Title: Usefulness and Predictive Capacity of ANI and SPI of the Hemodynamic Response to Standardized Stimuli During Neuro- and Urologic Surgery Under Standard Target Controlled Infusion of Propofol and Sufentanil.
Brief Title: Usefulness and Predictive Capacity of ANI and SPI of the Hemodynamic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veerle Van Mossevelde, Data Nurse, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ANI
Record Dates: First submitted 2015-11-05; First posted 2015-11-20 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Pain; Tachycardia; Hypertension
Keywords: ANI; SPI; Autonomic balance; Nociception measurement
MeSH Terms: conditions — Pain; Tachycardia; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metrodoloris Medical System (Experimental): Application of a skin electrode
  Interventions: Device: Metrodoloris Medical System; Device: Aisys® care station, Acertys
- Aisys® care station, Acertys (Active Comparator): SPI calculated from photoplethysmography
  Interventions: Device: Metrodoloris Medical System; Device: Aisys® care station, Acertys

INTERVENTIONS:
Device: Metrodoloris Medical System — Application of a skin electrode
  Other Names: ANI monitor
Device: Aisys® care station, Acertys — Standard photoplethysmography
  Other Names: SPI monitor

SUMMARY:
The primary objective of this study is to investigate the influence of a standardized noxious stimulus on the ANI, SPI and hemodynamic parameters during standard propofol and sufentanil TCI and to see if the ANI and SPI are predictive of a hemodynamic reaction.

In addition the investigators compare the performance of ANI and SPI against one another as well as investigate if ANI or SPI can be used to find the ideal CeSUF for a given patient.

DETAILED DESCRIPTION:
During general anesthesia hypnosis can be monitored routinely using EEG derivates like Bispectral index (BIS), entropy,.… However, monitoring analgesia or more precisely the nociceptive-antinociceptive (analgetic) balance during anesthesia proved more difficult. Clinical signs such as heart rate (tachycardia) or blood pressure (hypertension) are usually observed and used to assess nociception and a patient's autonomic unbalance. During general anesthesia administration of opioids like sufentanil and remifentanil decrease the ANS reactivity to noxious stimulation. Recently two variables based on standard anesthesia monitor equipment have been introduced into clinical practice: the Analgesia Nociception Index (ANI), derived from analysis of the small beat-to-beat oscillations of the heart rate during respiration, the heart rate variability (HRV), and the Surgical Pleth Index (SPI), calculated from the plethysmographic amplitude and heart beat interval.

ELIGIBILITY:
Inclusion Criteria:

* Male
* non-pregnant female participants
* ASA II-III
* >18-65 years
* Weight not exceeding 30% under or above ideal body weight
* Elective intracranial surgery or circumcision.

Exclusion Criteria:

* Use concurrent opioid containing drugs
* Use of any autonomic nervous system altering drugs
* History of opioid or alcohol abuse
* Hepatic, renal, metabolic, neuromuscular or cardiovascular disease
* Known allergies to anesthestetic / analgesic drugs
* Use of a peripheral nerve block, penile block

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The influence of a standardized noxious stimulus on pain measurement by means of analgesia nociception index (numerical score 0-100) | 30 minutes
  dimensionless number

SECONDARY OUTCOMES:
Predictive capacity of ANI and SPI of hemodynamic reactivity by means of analgesia nociception index (numerical score 0-100) or by SPI (numerical index 100-0) | 30 minutes
  Comparing the ANI and SPI before and during possible hemodynamic reactivity

CONTACTS AND LOCATIONS:
Overall Officials: Stef Cornelis, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Caroline Vanlersberghe, MD, Study Director — Universitair Ziekenhuis Brussel; Jan Poelaert, Prof. MD, Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Jette, Belgium